CLINICAL TRIAL: NCT06694961
Title: Knowledge of Adolescent Well-care Visits and Attitudes Amongst Pediatricians and Family Medicine Physicians Across Al-Ain City
Brief Title: Knowledge of Adolescent Well-care Visits and Attitudes Amongst Physicians
Status: Enrolling by invitation | Type: Observational
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Principal Investigator, Alaa Sattar Mehair, Pediatric Resident, Abu Dhabi Health Services Company
Other Study IDs: SEHA_Tawam-IRB KD/AJ/1072
Record Dates: First submitted 2024-11-04; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Health
Keywords: knowledge; Attitude; Pediatricians; family medicine; Physician; Adolescent; well-care visits
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Online Educational Material — Online educational material will be an easy way to reach large number of physicians

SUMMARY:
The goal of this observational study is to be a quality improvement project to assess the knowledge, attitude towards adolescent well visit screening and preventing counseling amongst pediatrician and family medicine physicians in Al-Ain city. We will be conducting an online survey covering general aspects regarding adolescent well-being visits, before and after providing necessary education to the participants

DETAILED DESCRIPTION:
This is a quality improvement project with the following fields to be studied:

* Knowledge of recommendations regarding adolescent well-care visits amongst pediatricians & primary care physicians in Al-Ain City.
* Compliance of pediatricians & primary care physicians towards adolescent well-care visits.
* Effectiveness in conducting educatory sessions for physicians to improve the quality of adolescent well-care visits.
* Adolescent behaviour & knowledge of the availability of well-care visits.
* Adolescent & family satisfaction in attendance of well-care visits.
* An online survey covering general aspects regarding adolescent well-being visits will be shared with pediatricians and family medicine physicians, before and after providing necessary education to the participants.

ELIGIBILITY:
Inclusion Criteria:

* Pediatricians and family medicine physicians at Al Ain City SEHA Hospitals.

Exclusion Criteria:

* Pediatricians and family medicine physicians who are not part of Al Ain City SEHA Hospitals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatricians and family medicine physicians
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge of physicians towards adolescent well care visits | 1 year
  The study will assess various aspects of physician's knowledge towards adolescents care including the required anticipatory guidance based on age including the Bright Futures Guidelines as per the American Academy of Pediatrics recommended screening and investigations through an online qualitative survey. The survey had 36 questions, with a mix of knowledge-based multiple choice questions and opinion questions ranging from strongly agree, agree, neutral, disagree, and strongly disagree.
Attitudes of physicians towards adolescent well-care visits | 1 year
  This study aims to highlight the attitude of pediatricians and family medicine physicians towards approaching adolescents for well-care visits. The survey had 36 questions, with a mix of knowledge-based multiple choice questions and opinion questions ranging from strongly agree, agree, neutral, disagree, and strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa S Mehair, MD, Principal Investigator — Abu Dhabi Health Services Co. -SEHA; Najla S AlKuawiti, MD, Study Chair — Abu Dhabi Health Services Co-SEHA
Locations (1):
- Tawam Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Bright Futures: Guidelines for Health Supervision of Infants, Children, and Adolescents, 4th Edition — https://www.aap.org/en/practice-management/bright-futures/bright-futures-materials-and-tools/bright-futures-guidelines-and-pocket-guide/